CLINICAL TRIAL: NCT01928498
Title: Evaluation of Drug Eluting Balloon for the Prevention of Hemodialysis Access Restenosis: A Prospective Randomized Trial (DEB Study)
Brief Title: Drug Eluting Balloon for Prevention of Hemodialysis Access Restenosis
Acronym: DEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Biotronik Canada Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE13.093 (2014-5032)
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Arteriovenous Fistulae; Arteriovenous Graft
Keywords: arteriovenous fistulae; arteriovenous graft; restenosis; angioplasty; drug eluting balloon
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel Eluting Balloon (Experimental): Paclitaxel Eluting Balloon Angioplasty
  Interventions: Device: Paclitaxel Eluting Balloon Angioplasty
- Conventional uncoated balloon (Active Comparator): Percutaneous Transluminal Angioplasty (PTA)
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA)

INTERVENTIONS:
Device: Paclitaxel Eluting Balloon Angioplasty
  Other Names: Passeo-18 Lux
  Arms: Paclitaxel Eluting Balloon
Device: Percutaneous Transluminal Angioplasty (PTA)
  Other Names: Passeo-18
  Arms: Conventional uncoated balloon

SUMMARY:
The purpose of this study is to evaluate the effectiveness of paclitaxel-coated balloon catheter to prevent restenosis after PTA (percutaneous transluminal angioplasty) of hemodialysis access (HA) in comparison with the uncoated PTA balloon catheter.

DETAILED DESCRIPTION:
In Canada, there are over 20,000 patients with chronic end-stage renal disease (ESRD)on long-term hemodialysis and the number is increasing rapidly.The creation of hemodialysis access (HA) (also called "lifeline" for dialysis patients) has become the most common type of vascular surgery. These HA are frequently complicated by dysfunction after their creation mainly due to neointimal hyperplastic stenosis (> 60% at one year). PTA is an established cornerstone method of treating stenotic lesions because of its minimally invasive percutaneous nature and widespread availability.Although PTA has a high initial success rate,narrowing will often recur in 2-3 months hence requiring further interventions. There are currently no durable therapies for the prevention or treatment of HA dysfunction restenosis after PTA.

Recently drug eluting balloon (DEB) with paclitaxel have repeatedly demonstrated their effectiveness to prevent restenosis due to intimal proliferation in the coronary and peripheral arterial systems. The investigators believe that the DEB with paclitaxel will significantly decrease the HA restenosis rate at the treated site and therefore will improve the management of HA failures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or hemodynamic evidence of HA dysfunction according to the clinician's judgment
* Patients with AVF (arteriovenous fistulae)or AVG (arteriovenous graft) located in the forearm or upper arm and is > 3 months old
* Minimum age of 18 years and written informed consent
* Target lesion stenosis is <3.0 cm in length and >50% in luminal diameter reduction
* Maximum of two secondary lesions (stenoses) if the following criteria are satisfied: The secondary lesion is located in the graft or peripheral veins, the secondary lesion is <3.0 cm in length and located >1.0 cm away from the target lesion, the secondary lesion is >50% luminal reduction compared to the reference vessel diameter
* Reference vessel diameter between 4 to 7 mm
* The HA must not be thrombosed and the lesion can be crossed with guide wire before angioplasty
* Lesion site: from 2 cm above the arterial anastomosis to the superior vena cava
* Restenotic lesion (previously treated by PTA or stent) or de novo lesion

Exclusion Criteria:

* Contraindication to angiography or PTA
* Intervention of the HA circuit within the past 30 days
* Systemic infection or a local infection associated with the graft
* The patient is pregnant
* Patient is enrolled in another investigational study.
* Life expectancy < 12 months
* History of severe allergic reaction to contrast media or to paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Late lumen loss (LLL) at 6 months after PTA (percutaneous transluminal angioplasty) | 6 months
  Comparison of the mean LLL (late lumen loss) in patients in the two trial arms (DEB vs plain PTA) evaluated by quantitative angiography at six months after PTA.
  LLL is defined as the difference between the MLD (minimum lumen diameter) immediately after balloon angioplasty and the MLD at follow-up

SECONDARY OUTCOMES:
The angiographic percentage of diameter stenosis and the incidence of angiographic binary restenosis rate (≥50% of the diameter of the reference-vessel segment) | 6 months
  The change in the degree of stenosis (in %) at the intervention site between the measure right after the intervention, and 6 months later and the difference between restenosis rates in the two trial arms at 6 months.
Change of HA flow | Before angioplasty, week 1, month 1or month 3
  Difference between mean HA flow in the two groups (measured at the same times)
The rate of HA failure | 3 months
  Time elapsed from the initial intervention (at randomization) to the earliest (if any) of these 3 events: HA thrombosis, HA re-intervention (surgical or endovascular, including creation of a new HA), or CVC (central venous catheter) insertion for dialysis purpose
Drug eluting balloon safety | 3 months
  Proportion of patients with side effects in the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Éric Therasse, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (3):
- Canada (3):
  - Hôpital Charles-Lemoyne, Longueuil, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'université de Montréal-CHUM, Montreal, Quebec